CLINICAL TRIAL: NCT06669611
Title: Nab-TPC Versus GP Chemotherapy Combined With Camrelizumab in the Treatment of Recurrent/Metastatic Nasopharyngeal Carcinoma: Randomized Controlled, Multi Center, Phase III Clinical Study
Brief Title: Nab-TPC vs GP Combined With Camrelizumab in the Treatment of Recurrent/Metastatic Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, XIANG YANQUN, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2024-869-01
Record Dates: First submitted 2024-10-29; First posted 2024-11-01 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Nasopharyngeal Cancinoma (NPC)
MeSH Terms: interventions — camrelizumab; Cisplatin; Gemcitabine; 130-nm albumin-bound paclitaxel; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Camrelizumab with GP chemotherapy (Active Comparator): Camrelizumab, cisplatin and gemcitabine
  Interventions: Drug: Camrelizumab combined GP chemotherapy
- camrelizumab with nab-TPC chemotherapy (Experimental): camrelizumab plus nab-TPC chemotherapy (nab-paclitaxel, cisplatin and capecitabine)
  Interventions: Drug: Camrelizumab combined TPC chemotherapy

INTERVENTIONS:
Drug: Camrelizumab combined GP chemotherapy — Camrelizumab was intravenously given at dose of 200 mg on day 1. The GP regimen included gemcitabine administered at a dose of 1 g/m2 on day 1 and day 8, cisplatin at a dose of 80 mg/m2 on day 1.Q3W 1 cycle, 4-6 cycles.
  Other Names: Camrelizumab, cisplatin and gemcitabine
  Arms: Camrelizumab with GP chemotherapy
Drug: Camrelizumab combined TPC chemotherapy — Camrelizumab was intravenously given at dose of 200 mg on day 1. The TPC regimen included nab-paclitaxel administered at a dose of 200 mg/m2 on day 1, cisplatin at a dose of 60 mg/m2 on day 1, and capecitabine at a dose of 1000 mg/m2, taken orally twice a day on days 1 to 14, for each cycle. Q3W 1 cycle, 4-6 cycles.
  Other Names: camrelizumab plus nab-TPC chemotherapy, nab-paclitaxel, cisplatin and capecitabine
  Arms: camrelizumab with nab-TPC chemotherapy

SUMMARY:
We expect to conduct a clinical trial in recurrent and metastatic nasopharyngeal carcinoma patients to explore and compare the efficacy and safety of induction chemotherapy (TPC vs. GP) with combination therapy of Camrelizumab.

DETAILED DESCRIPTION:
The therapeutic effect of patients with metastatic nasopharyngeal carcinoma has been further improved. Numerous previous studies have shown that anti-PD-1 immune checkpoint inhibitors (ICIs) have strong activity in treated metastatic nasopharyngeal carcinoma patients, with an objective response rate (ORR) of 20-34%. In addition, immunotherapy has also achieved good results in the first-line treatment of recurrent/metastatic nasopharyngeal carcinoma. In 2021, the clinical results of a study on the treatment of recurrent/metastatic nasopharyngeal carcinoma with pembrolizumab were published. The median PFS of the pembrolizumab combined with chemotherapy group was 9.7 months, significantly prolonging PFS, with an HR value of 0.54, and reducing the risk of disease progression by 46%. Based on this, the 2022 CSCO guidelines will use pembrolizumab combined with GP chemotherapy as a new first-line treatment for metastatic nasopharyngeal carcinoma.We conducted a study comparing the efficacy of GP regimen and nab TPC regimen, and found that nab TPC regimen significantly improved the survival of patients with metastatic nasopharyngeal carcinoma compared to GP regimen, and the nab TPC regimen group had milder grade 3-4 toxic side effects.This study aims to design a prospective phase III clinical trial on the safety and efficacy of GP combined with Carilizumab compared to nab TPC regimen combined with Carilizumab chemotherapy for recurrent and metastatic nasopharyngeal carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years.
2. ECOG score of 0-1.
3. Expected survival of at least 12 weeks.
4. Recurrent/Metastatic Nasopharyngeal Carcinoma.
5. At least 4 weeks since the previous chemotherapy.
6. At least one (according to RECIST) measurable lesion, lesions that have been previously irradiated can not be considered target lesions.
7. had adequate organ function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2027-11-20 (Estimated); Study Completion 2029-11-20 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | 15 months
  The primary endpoint was PFS, which was assessed as the time from randomization to disease progression per RECIST v1.1 assessed by IRC or death, whichever occurred first.

SECONDARY OUTCOMES:
Overall Survival | 1,3,5 years
  The secondary endpoint was OS, which was assessed as the time from randomization to death according to RECIST v1.1 or PERCIST, whichever occurred first.
Safety and Adverse Events | 3 months
  Adverse events occurring during chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- SunYat-senU, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No